CLINICAL TRIAL: NCT06563297
Title: To Explore the Optimal Dose of Alfentanil for Skull Pin Fixation Under Surgical Pleth Index Monitor in Intracranial Surgery
Brief Title: To Explore the Optimal Dose of Alfentanil for Skull Pin Fixation in Intracranial Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KMUHIRB-F(II)-20240191
Record Dates: First submitted 2024-08-18; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-06

CONDITIONS: Procedural Pain
Keywords: alfentanil; pain; surgical pleth index
MeSH Terms: conditions — Pain, Procedural; Pain | interventions — Alfentanil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant Group (Experimental): Neurosurgery with fixation
  Interventions: Drug: Alfentanil

INTERVENTIONS:
Drug: Alfentanil — We first start with alfentanil 100 ng/ml, and use the up and down method as adjust 25 ng/ml of concentration of alfentanil each time. An SPI higher than 80 and hyperdynamics (the increased HR and MBP up 20% of baseline or HR>100bpm and ABP>180/100mmHg) indicates insufficient analgesia, therefore increase it by 25 ng/ml at the next patient; an SPI lower than 80 and stable hemodynamics (the changes of HR and MBP within 20% of baseline or HR<50bpm and ABP<90/50mmHg) indicates that analgesia is acceptable, and the next patient will decrease it by 25 ng/ml during skull pin fixation. If the analgesia is inadequate, increase alfentanil concentration will be prescribed. On the other hand, if analgesia is adequate, however hyperdynamics was noted, beta blocker or calcium channel blocker will be prescribed. If hypotension (ABP<90/50 mmHg) or bradycardia (HR<50 bpm) occur, we first stop alfentanil infusion and treated with ephedrine or atropine, respectively.

SUMMARY:
Forty patients were enrolled, and all patients used total intravenous anesthesia (alfentanil-propofol based TIVA) as anesthesia induction and maintenance. According to our experience, patients who underwent intracranial surgery for skull pin fixation used alfentanil 100 ng/ml, while the hemodynamics is relatively stable. Therefore, when this plan is implemented, the patient needs to be under the same depth of anesthesia (monitored by EEG, maintaining a value of 40-60), first start with alfentanil 100 ng/ml, and use the up and down method as adjust 25 ng/ml of concentration of alfentanil each time. An SPI higher than 80 and hyperdynamics (the increased HR and MBP up 20% of baseline or HR>100bpm and ABP>180/100mmHg) indicates insufficient analgesia, therefore increase it by 25 ng/ml at the next patient; an SPI lower than 80 and stable hemodynamics (the changes of HR and MBP within 20% of baseline or HR<50bpm and ABP<90/50mmHg) indicates that analgesia is acceptable, and the next patient will decrease it by 25 ng/ml during skull pin fixation. If the analgesia is inadequate, increase alfentanil concentration will be prescribed. On the other hand, if analgesia is adequate, however hyperdynamics was noted, beta blocker or calcium channel blocker will be prescribed. If hypotension (ABP<90/50 mmHg) or bradycardia (HR<50 bpm) occur, we first stop alfentanil infusion and treated with ephedrine or atropine, respectively.

Data collection: HR, MBP, SPI, BIS, systolic pressure variation (SPV), pulse pressure variation (PPV) , concentrations of propofol and alfentanil before 2 mins, during, 5, and 15 mins of skull pin fixation were recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years old and less than 80 years old
* With anesthesia risk grade below grade three (including grade three) (ASA I~III)
* Patients who are expected to undergo intracranial surgery for skull pin fixation

Exclusion Criteria:

* Those with anesthesia risk classification ASA class IV or higher
* Those who are allergic to alfentanil or propofol drugs
* Emergency patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-13 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
50% effect concentration of alfentanil | peri-fixation period
  50% effect concentration of alfentanil will be recorded at 2 mins before fixation, during fixation, 5 mins after fixation, and 15 mins after fixation.
95% effect concentration of alfentanil | peri-fixation period
  95% effect concentration of alfentanil will be recorded at 2 mins before fixation, during fixation, 5 mins after fixation, and 15 mins after fixation.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No